CLINICAL TRIAL: NCT06182462
Title: The Effects of A Virtual Reality Game on Anxiety During Dental Procedures in Children (VR-TOOTH): A Randomized, Controlled Trial Protocol
Brief Title: Virtual Reality Distraction for Dental Anxiety (RCT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VR-TOOTH - RCT
Record Dates: First submitted 2023-08-17; First posted 2023-12-27 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Dental Anxiety; Dental Phobia; Dental Trauma; Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Distraction (Experimental): Use of virtual reality (VR) during dental procedure.
  Interventions: Device: Virtual Reality Distraction
- Standard Treatment (Active Comparator): Dental Clinic's standard treatment during dental procedure.
  Interventions: Device: Dental Clinic's Standard Treatment

INTERVENTIONS:
Device: Virtual Reality Distraction — The experimental group will receive a VR video game called "DREAM DENTAL" designed specifically for this study. Pharmaceutical treatment during the procedure such as the use of injected local anesthesia will be used if the procedure requires. Children will be able to play for the entire duration of the dental procedure. The VR video game aims at reducing anxiety in children aged 6 to 17 years old by means of immersive distraction. The VR headset offers children with the ability of viewing the game they are playing in real time while simultaneously obstructing the partial view they would normally have of the procedure. In the event of non-cooperation during the appointment, any retake or re-scheduling appointments will be compiled by the research assistant or resident dentist. One parent will be allowed in the room during the dental procedure and their presence will be recorded.
  Arms: Virtual Reality Distraction
Device: Dental Clinic's Standard Treatment — The control group will only receive a care-as-usual approach. This includes viewing cartoons on a muted mounted television set and the use of pharmaceutical treatment during the procedure such as the use of injected local anesthesia, according to the procedure. In the event of non-cooperation during the appointment, any retake or re-scheduling appointments will be compiled by the research assistant. One parent will be permitted to be present in the room during the procedure as part of the clinic's usual protocol and their presence will be recorded. Children allocated to the control group will be offered the possibility to try the VR game after the study period if they choose to do so.
  Arms: Standard Treatment

SUMMARY:
The aim of this randomized clinical trial is to verify the efficacy of VR immersion over a muted cartoon on a wall-mounted TV to decrease dental fear and anxiety of children undergoing dental procedures. The study also aims to gain insight on the satisfaction of parents and healthcare providers on the use of VR during dental appointments.

Main research question: Does VR immersion compare to a cartoon on a wall-mounted TV is more efficacious to decrease dental fear and anxiety of children requiring dental procedures?

Participants will be playing through a VR immersive game wearing a eye-tracking VR headset that requires no movement of the head to play, facilitating the dental procedure.

The investigators will take measures of the stress levels of participants and their parents using a validated stress scale and also by taking salivary samples to verify the levels of a stress biomarker (alpha-amylase).

DETAILED DESCRIPTION:
Background

Dental fear and anxiety (DFA) is a condition that affects approximately 13.3% to 29.3% of children and adolescents, and is a significant cause of patients avoiding dental care. In children, DFA is also associated with a lower oral-health-related quality of life. Although the etiology of DFA is multifactorial, a previous traumatic dental experience is the most predictive factor for DFA. The majority of DFA experienced by adults stems from poor dental experiences as children. Short term distress during appointments that is not managed properly can accumulate into poor dental experiences, and in turn, reinforcing DFA into adulthood.

Dental patients with special health care needs (SHCN) are defined as patients requiring additional time and special consideration when receiving treatment due to medical, physical, cognitive or developmental conditions. The population includes children with behaviour (e.g. autism spectrum, anxiety, ADHD), congenital (e.g. trisomy 21, congenital heart disease), developmental (e.g. cerebral palsy), systemic (e.g. childhood cancer, sickle cell disease), or cognitive disorders (eg. intellectual disability). Children with SHCN face more barriers to dental care than the overall population. Barriers include external factors (transportation, cost, inadequate dental facilities) and internal factors (fear and poor tolerance). Many children with SHCN are cared for by dentists in the community, or more often times, in hospital dental clinic settings. They likewise experience more anxiety than those without a disability, which can result in more difficult dental visits or multiple reports of visits.

Understanding and assessing DFA in children is important for delivering successful dental care with high satisfaction in this age group. Among the vast assessment method options available today, self-report assessment, parental proxy assessment, observation-based assessment and physiological assessment are the four major types of measures for children with SHCN. Further, salivary alpha-amylase, an enzyme correlated to both adrenaline and noradrenaline, has also been used as a biomarker for autonomic nervous system activity and stress.

Factors in the dental setting that trigger DFA include the loud sounds of dental instruments, presence of strangers examining the oral cavity, and the fear of pain. Of these, the anticipation and use of local anesthetic injections are by far the main triggers. Although necessary to provide adequate pain control during certain treatments, local anesthetic injections are uncomfortable. For children, the initial injection combined with the feeling of numbness during the procedure is especially distressing. Pharmacological agents, combined with light to moderate sedation, or general anesthesia can also be considered for non-cooperative patients, but they are often time consuming and at a higher cost as well as generating health risks. Audiovisual distractions such as tablets/TV screens have been used as distraction techniques during dental procedures with overall positive results. However, there is a lack of interactivity of these techniques, and as a result, are not enough to distract children from the stressful procedure. Further, lack of patient cooperation due to DFA often requires dentists treating pediatric populations to end appointments prematurely, and sometimes without completion of the planned procedure. Treating an anxious and fearful patient can also create an environment of stress for the clinician and associated dental team.

Moreover, when treating children with SHCN, extra time and tools are needed to provide comfortable dental care. Depending on the child's diagnosis, many have hypersensitivity to external stimuli such as loud noises, aversion to specific tastes and difficultly straying from usual daily routines. A study by Pagano and colleagues showed that the use of augmented reality was well suited for patients with autism spectrum disorder in preparation for their dental visits. Additionally, a systematic review by Cunningham and colleagues concluded that virtual reality was a promising tool in dentistry, especially with the population of children with autism spectrum disorder or other special needs.

Aim of the Study

The aim of the study is to verify the efficacy of a VR immersion game compared to a muted cartoon on a wall-mounted TV, to decrease anxiety in pediatric special needs patients undergoing dental procedures. The study also aims to gain insight on parent and healthcare providers' satisfaction levels on the use of VR during dental appointments.

Objectives

The primary research objective is to determine:

1. The efficacy of a VR immersion game to decrease dental fear and anxiety in children with special needs requiring dental procedures compared to the standard intervention consisting of watching a cartoon on a muted mounted-TV set.

The secondary objectives of this study are as follows:

1. To compare parents' and healthcare professionals' satisfaction levels between the VR distraction group and the standard intervention group.
2. To compare physiological parameters (pulse, oxygen saturation and salivary alpha-amylase) between the VR distraction group and the standard intervention group.
3. To compare the occurrence of side effects between the VR distraction group and the standard intervention group.
4. To compare dental procedure length between the VR distraction group and the standard intervention group.
5. To compare the rate of dental procedures' completion between the VR distraction group and the standard intervention group.

MATERIALS AND METHODS

Design This randomized controlled trial study will follow a parallel design including two groups: a control group (watching cartoons on a muted mounted wall TV set) and an experimental group (virtual reality game during the dental procedure).

Sample and Setting

This study will include 88 participants including an attrition rate of 10%. All participants in this study will be allocated in an equal ratio of 44 per group. Recruitment will be carried out at the dental clinic of the Centre Hospitalier Universitaire Sainte-Justine, a pediatric hospital in Montréal, Canada. This clinic mostly serves patients with special health care needs such as craniofacial abnormalities, autism spectrum disorder, children battling cancer, and others. Pediatric patients with SHCN represent around 80% of the total clientele of this clinic while the rest is comprised of otherwise healthy patients with dental traumas and other dental emergencies. Participants will be identified by the clinic's resident dentist using the scheduling system for upcoming appointments for specific painful dental procedures such as teeth extractions, fillings, and others. The research assistants will proceed to contact the parents or legal guardian in order to provide information on the study and seek parents' approval ahead of time. An individual independent of the clinical dental will review consent with participants and their parents. The information and consent form will be signed by one of the parents on the day of the visit.

Randomization and allocation

Randomization will be done through the electronic RedCap system. Allocation to either intervention will be randomized by an independent biostatistician from the URCA (Applied Clinical Research Unit). In order to equalize participants in both arms, permuted block randomization with randomly selected block sizes design will be used to randomize participants to their intervention. Access to the randomization list will only be granted to the biostatistician and allocation will be concealed using RedCap (Research Electronic Data Capture) to reduce selection bias.

Measure of primary outcome

DFA scores will be evaluated using the Venham Anxiety and Behavioral Scale. It is an observation-based assessment by proxy for dental fear and anxiety and are among the most frequent behavior scoring models for DFA. It is composed of two scales used to assess the anxiety and uncooperative behavior of children in the dental setting. The scale is also found under the name Clinical Anxiety Scale/Uncooperative Behaviour Rating Scale (CARS/BRS) or Venham Clinical Cooperation Scale (VCCS) and Venham Clinical Anxiety Scale (VCAS) and has been used as anxiety rating scale in other studies that evaluate the efficacy of VR distraction in the management of DFA . Both scales consist of a 6-point scale, with 6 defined behavioral levels that range from 0 to 5. The highest score defines the highest anxiety level or lack of cooperation. A high degree of reliability is seen for both scales, even for untrained observers . The scale points are measured by proxy and anchored in objective, specific, and readily observable behaviors. The research assistant will evaluate the participant's behavior by picking a number from 0 to 5 according to the scale, thus for each participant, two scores on the levels of anxiety and cooperation for the dental procedure will be obtained at T0, T1 and T2. These scores will also be validated and allocated as a consensus with the attending dentist or dental professional. Venham and colleagues pointed out that the scale is reliable and valid and provides interval level measurement. It is demonstrated that the scale is proven as a useful instrument for assessing child's responses to dental stress. Anxiety score and uncooperative score will both be evaluated at T0 (baseline), during the procedure at 10 minutes after the beginning of the procedure (T1) or at mid-procedure for shorter dental treatments, and after the completion of the procedure (T2).

Virtual reality and Game Specification

Virtual reality (VR) is defined as an artificial environment which is experienced through sensory stimuli. It is a modern tool that can immerse patients in a "game" or "world." Commonly used in the medical field to help distract patients during unpleasant procedures such as vaccination and cast removal, it has proven to be effective at decreasing anxiety and providing a more positive experience for patients. A recent clinical trial by Alshatrat and colleagues concluded that VR is an effective tool in reducing anxiety in young children during dental procedures. Moreover, a previous study by Ram and colleagues showed that both parent and clinician satisfaction was high using audio-visual glasses as distraction for children during dental treatments. However, clinical VR research in pediatric dentistry is limited, especially with special needs populations. VR use in pediatric dentistry offers the potential of an additional non-pharmacologic tool.

Developed by Paperplane Therapeutics, "DREAM DENTAL" is tailored for the pediatric population and approved by a team of healthcare professionals in pediatric care. The simplified no-success game allows it to be enjoyable no matter the child's video game experience. It was designed specifically for this study with the specific horizontal position in mind needed for dental procedures. The video game is designed to be supported by the Pico Neo 4 VR headset.

The objective of the VR game is to shoot lasers at targets located on the islands, such as balloons and trolls. It uses a new eye-tracking technology developed within the headset to help direct laser beams without any head movement, making it easier for dental procedures where head movement is restricted. These features also aim to reduce cybersickness. The preliminary version of the VR headset has been tested in clinic on staff - the size and volume of the headset do not hinder delivery of dental care, but this will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 to 17 years;
2. Received the dentist's recommendation to participate;
3. Required to undergo any dental procedure;
4. Accompanied by a parent or a legal guardian who can understand, read, and write in either French or English.

Exclusion Criteria:

1. Suffer from epilepsy,
2. Paralysis or paresis of the hand
3. Has any diagnosed eye disease/problem,
4. Any other conditions preventing them from using virtual reality (VR) (e.g., epidermolysis bullosa).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Anxiety scale score is recorded by the operator at the following timepoints: Before the dental procedure to establish baseline; immediately after the completion of dental intervention appointment
  To evaluate and observe preliminary effects of VR distraction, we will be using the Venham Anxiety and Behavioural Scale (VABRS). It is an observation-based assessment by proxy for dental fear and anxiety and are among the most frequent behavior scoring models for DFA. It is composed of two scales used to assess the anxiety and uncooperative behavior of children in the dental setting. Both scales consist of a 6-point scale, with 6 defined behavioral levels that range from 0 to 5. The highest score defines the highest anxiety level or lack of cooperation.

SECONDARY OUTCOMES:
Parent's or legal guardian satisfaction | Satisfaction questionnaire is reported by parents immediately following completion of the dental procedure
  Parent's or legal guardian's satisfaction on the intervention and side effects will be assessed using the Visual analog Scale, (0-10, where 0 is very dissatisfied and 10 in very satisfied) and following the recommended question by Pediatric Initiatives on Methods, Measurement and Pain Assessment in Clinical Trials (PedIMMPACT): "Considering anxiety relief, side effects and emotional recovery, how satisfied were you with the intervention used to manage anxiety experienced by your child?"
Healthcare professional's satisfaction | Satisfaction questionnaire is reported by healthcare professional immediately following completion of the dental procedure
  Healthcare professional's satisfaction on the intervention will be assessed using the Visual Analog Scale, (VAS; ranked from 0-10, where 0 is very dissatisfied and 10 in very satisfied) as well as a 6-question satisfaction questionnaire (each answer will be given a score of 1,2,3,or 4 based on the choice of response (respectively: Totally disagree, Disagree, Agree, Totally agree) and will result in a final score between 6 and 24.
Heart rate in beats per minute | Heart rate will be measured immediately before the procedure and for the entire duration of the procedure (Approximately 30-60 minutes)
  Heart rate will be continuously measured using COVIDIEN Nellcor psaturation meter, an approved and validated device.
Oxygen saturation | Oxygen saturation will be measured immediately before the procedure and for the entire duration of the prodedure (Approximately 30-60 minutes)
  Oxygen saturation will be continuously measured using COVIDIEN Nellcor pulse oxygen saturation meter, an approved and validated device.
Salivary alpha-amylase | Salivary Alpha-Amylase will be measured immediately before and 10-minutes after the procedure
  Salivary alpha-amylase will be taken to quantify stress level
Occurrence of side effects | Any side effects will be noted along with the time at which they occurred during the procedure.
  Occurrence of side effects will be collected from arrival on site to discharge from study using a checklist of common side effects experienced by children in both groups while using VR and also related to dental medication.
Length of procedure in minutes | Reported immediately after the procedure.
  Length of procedure will be measured and collected for every participant and compared to average duration for similar procedure that will have been measured prior to the study by the clinic's personnel.
Intervention completion | Intervention completion will also be documented by the research assistant at the end of the dental procedure.
  To compare the intervention completion due to DFA between the VR distraction group and the standard intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- St.Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cianetti S, Lombardo G, Lupatelli E, Pagano S, Abraha I, Montedori A, Caruso S, Gatto R, De Giorgio S, Salvato R. Dental fear/anxiety among children and adolescents. A systematic review. Eur J Paediatr Dent. 2017 Jun;18(2):121-130. doi: 10.23804/ejpd.2017.18.02.07. PMID 28598183
- [Background] Murad MH, Ingle NA, Assery MK. Evaluating factors associated with fear and anxiety to dental treatment-A systematic review. J Family Med Prim Care. 2020 Sep 30;9(9):4530-4535. doi: 10.4103/jfmpc.jfmpc_607_20. eCollection 2020 Sep. PMID 33209758
- [Background] Luoto A, Lahti S, Nevanpera T, Tolvanen M, Locker D. Oral-health-related quality of life among children with and without dental fear. Int J Paediatr Dent. 2009 Mar;19(2):115-20. doi: 10.1111/j.1365-263X.2008.00943.x. PMID 19250394
- [Background] Beaton L, Freeman R, Humphris G. Why are people afraid of the dentist? Observations and explanations. Med Princ Pract. 2014;23(4):295-301. doi: 10.1159/000357223. Epub 2013 Dec 20. PMID 24356305
- [Background] Humphris G, King K. The prevalence of dental anxiety across previous distressing experiences. J Anxiety Disord. 2011 Mar;25(2):232-6. doi: 10.1016/j.janxdis.2010.09.007. Epub 2010 Sep 19. PMID 20952156
- [Background] Ten Berge M, Veerkamp JS, Hoogstraten J. The etiology of childhood dental fear: the role of dental and conditioning experiences. J Anxiety Disord. 2002;16(3):321-9. doi: 10.1016/s0887-6185(02)00103-2. PMID 12214817
- [Background] Shim YS, Kim AH, Jeon EY, An SY. Dental fear & anxiety and dental pain in children and adolescents; a systemic review. J Dent Anesth Pain Med. 2015 Jun;15(2):53-61. doi: 10.17245/jdapm.2015.15.2.53. Epub 2015 Jun 30. PMID 28879259
- [Background] Oliveira MA, Vale MP, Bendo CB, Paiva SM, Serra-Negra JM. Influence of negative dental experiences in childhood on the development of dental fear in adulthood: a case-control study. J Oral Rehabil. 2017 Jun;44(6):434-441. doi: 10.1111/joor.12513. Epub 2017 May 3. PMID 28386938
- [Background] Koneru A, Sigal MJ. Access to dental care for persons with developmental disabilities in Ontario. J Can Dent Assoc. 2009 Mar;75(2):121. PMID 19267962
- [Background] Yon MJY, Chen KJ, Gao SS, Duangthip D, Lo ECM, Chu CH. An Introduction to Assessing Dental Fear and Anxiety in Children. Healthcare (Basel). 2020 Apr 4;8(2):86. doi: 10.3390/healthcare8020086. PMID 32260395
- [Background] Vacaru RP, Didilescu AC, Sfeatcu R, Tanase M, Munteanu A, Miricescu D, Kaman WE, Brand HS. The Effect of Dental Treatments in Caries Management on Stress and Salivary Protein Levels. J Clin Med. 2022 Jul 27;11(15):4350. doi: 10.3390/jcm11154350. PMID 35893440
- [Background] Morgan AG, Rodd HD, Porritt JM, Baker SR, Creswell C, Newton T, Williams C, Marshman Z. Children's experiences of dental anxiety. Int J Paediatr Dent. 2017 Mar;27(2):87-97. doi: 10.1111/ipd.12238. Epub 2016 Jul 4. PMID 27376925
- [Background] Al-Khotani A, Bello LA, Christidis N. Effects of audiovisual distraction on children's behaviour during dental treatment: a randomized controlled clinical trial. Acta Odontol Scand. 2016 Aug;74(6):494-501. doi: 10.1080/00016357.2016.1206211. Epub 2016 Jul 13. PMID 27409593
- [Background] Alshatrat SM, Sabarini JM, Hammouri HM, Al-Bakri IA, Al-Omari WM. Effect of immersive virtual reality on pain in different dental procedures in children: A pilot study. Int J Paediatr Dent. 2022 Mar;32(2):264-272. doi: 10.1111/ipd.12851. Epub 2021 Jul 5. PMID 34133809
- [Background] Pagano S, Lombardo G, Coniglio M, Donnari S, Canonico V, Antonini C, Lomurno G, Cianetti S. Autism spectrum disorder and paediatric dentistry: A narrative overview of intervention strategy and introduction of an innovative technological intervention method. Eur J Paediatr Dent. 2022 Mar;23(1):54-60. doi: 10.23804/ejpd.2022.23.01.10. PMID 35274543
- [Background] Cunningham A, McPolin O, Fallis R, Coyle C, Best P, McKenna G. A systematic review of the use of virtual reality or dental smartphone applications as interventions for management of paediatric dental anxiety. BMC Oral Health. 2021 May 7;21(1):244. doi: 10.1186/s12903-021-01602-3. PMID 33962624
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Ram D, Shapira J, Holan G, Magora F, Cohen S, Davidovich E. Audiovisual video eyeglass distraction during dental treatment in children. Quintessence Int. 2010 Sep;41(8):673-679. PMID 20657857
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Venham LL. The effect of mother's presence of child's response to dental treatment. ASDC J Dent Child. 1979 May-Jun;46(3):219-25. No abstract available. PMID 285948
- [Background] Sahebalam R, Rafieinezhad R, Boskabad M. Comparison of the Efficacy of Jilo Animation Approach versus Conventional Tell-Show-Do (TSD) Technique on Cooperation and Anxiety Levels of Children during Dental Practice: A Randomized Controlled Clinical Trials. J Dent (Shiraz). 2020 Dec;21(4):284-291. doi: 10.30476/dentjods.2020.81897.1001. PMID 33344678
- [Background] Nunna M, Dasaraju RK, Kamatham R, Mallineni SK, Nuvvula S. Comparative evaluation of virtual reality distraction and counter-stimulation on dental anxiety and pain perception in children. J Dent Anesth Pain Med. 2019 Oct;19(5):277-288. doi: 10.17245/jdapm.2019.19.5.277. Epub 2019 Oct 30. PMID 31723668
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251
- [Background] Furlan NF, Gaviao MB, Barbosa TS, Nicolau J, Castelo PM. Salivary cortisol, alpha-amylase and heart rate variation in response to dental treatment in children. J Clin Pediatr Dent. 2012 Fall;37(1):83-7. doi: 10.17796/jcpd.37.1.n32m21n08417v363. PMID 23342572
- [Background] Alaki SM, Safi A, Ouda S, Nadhreen A. Comparing Dental Stress in New Child Patients and Returning Patients Using Salivary Cortisol, Immunoglobulin-A and Alpha- Amylase. J Clin Pediatr Dent. 2017;41(6):462-466. doi: 10.17796/1053-4628-41.6.8. Epub 2017 Sep 22. PMID 28937902
- [Background] AlMaummar M, AlThabit HO, Pani S. The impact of dental treatment and age on salivary cortisol and alpha-amylase levels of patients with varying degrees of dental anxiety. BMC Oral Health. 2019 Sep 6;19(1):211. doi: 10.1186/s12903-019-0901-7. PMID 31492133
- [Background] Chaturvedi Y, Chaturvedy S, Marwah N, Chaturvedi S, Agarwal S, Agarwal N. Salivary Cortisol and Alpha-amylase-Biomarkers of Stress in Children undergoing Extraction: An in vivo Study. Int J Clin Pediatr Dent. 2018 May-Jun;11(3):214-218. doi: 10.5005/jp-journals-10005-1514. Epub 2018 Jun 1. PMID 30131644